CLINICAL TRIAL: NCT04137172
Title: Short Term Outcomes of Laparoscopic Intraperitoneal Onlay Mesh With Facial Repair(IPOM-plus) for Ventral Hernia. A Randomized Controlled Trial
Brief Title: Short Term Outcomes of Laparoscopic Intraperitoneal Onlay Mesh With Facial Repair(IPOM-plus) for Ventral Hernia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, osama khalil, assistant profeosser, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR-17324-2
Record Dates: First submitted 2019-10-14; First posted 2019-10-23 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Hernia
Keywords: ventral hernia - LVHR-transfacial repair
MeSH Terms: conditions — Hernia | interventions — Laparoscopy; Herniorrhaphy; Wound Healing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group1 (Experimental): underwent laparoscopic IPOM hernioplasty without repair
  Interventions: Procedure: laparoscopic (IPOM) hernioplasty without repair
- group2 (Experimental): underwent laparoscopic IIPOM hernioplasty with intracorporeal repair using proline 0 versus stratifix PDS
  Interventions: Procedure: aparoscopic IIPOM hernioplasty with intracorporeal repair using proline 0 versus stratifix PDS
- group3 (Experimental): underwent laparoscopic IPOM hernioplasty with transfacial closure using PDS LOOP 0
  Interventions: Procedure: laparoscopic IPOM hernioplasty with transfacial closure using PDS LOOP 0

INTERVENTIONS:
Procedure: laparoscopic (IPOM) hernioplasty without repair — Under general anesthesia, supine position, lateral visiport 12mm was inserted at the left anterior axillary line . Other two 5mm ports were inserted under vision. A 30-degree optics were used. Adhesiolysis was done . The contents of hernia were reduced . The borders of the defect were illuminated and outlined. The abdominal wall was marked from outside for measurement of defect size and for corners fixation of mesh with 5cm away from defect edge. Defect with axis from 9 to 12 cm is considered big defect.
  Group I:
  Proline (1) sutures were applied at the corners of the mesh introduced into the peritoneal cavity. Endoclose passed at the marked site from abdominal wall, sutures hanged and tied subcutaneously, completion of mesh fixation using secure strap .
  Arms: group1
Procedure: aparoscopic IIPOM hernioplasty with intracorporeal repair using proline 0 versus stratifix PDS — Group II:
  Using PDS 0, a stratifix suture (STRATAFIX™ Symmetric PDS™ Plus Knotless Tissue Control Device) versus proline 1 , used to repair and plicate the defect then mesh fixation
  Arms: group2
Procedure: laparoscopic IPOM hernioplasty with transfacial closure using PDS LOOP 0 — The PDS loop sutures were prepared by cutting the needles, keeping two detached ends and one blind end. A small curved supraumbilical incision was done. The endoclose passed through upper border of incision penetrating the abdominal wall above the defect, hanging the blind end of the PDS Loop to outside. It passed through the lower border of the wound crossing the defect. It hanged one detached end of the PDS Loop suture to outside, passed again through lower border of incision to catch the other detached end. The two ends were hanged not tied to avoid incision closure. The process is repeated by passing 1-2 cm lateral or medial to the previous sutures, then blind ends were divided. Lastly, all sutures are tied. Mesh was fixed as before.
  Arms: group3

SUMMARY:
entral hernias are a major cause of functional impairment, abdominal pain, and bowel obstruction. The overall incidence of primary ventral hernia is estimated to be between 4 and 5 % in the literature, and ventral incisional hernia rates vary from 35 to 60 % within 5 years after laparotomy . After laparoscopy, this rate is estimated to decline from 0.5 to 15 % even after two decades, LVHR or open repair (OVHR) is still a matter of debate because of concerns about seroma formation, recurrence rate, and the intraperitoneal mesh position. . The laparoscopic technique for repairing ventral and incisional hernias is now well established. However, several issues related to LVHR, such as the high recurrence rate of hernias with large fascial defects and in extremely obese patients, are yet to be resolved. Additional problems include seroma formation. To solve these problems, laparoscopic fascial defect closure with IPOM reinforcement (IPOM-Plus) has been introduced in the past decade, and a few studies have reported satisfactory outcomes. Although detailed techniques for fascial defect closure and handling of the mesh have been published, standardized techniques are yet to be established.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years undergoing surgery for primary or incisional ventral hernia
* defect whose major axis not exceeding 12cm.

Exclusion Criteria:

* Patients undergoing revision
* Emergency surgery.
* Parastomal hernias were not included.
* Patients not candidate for laparoscopy including cardiac and COPD patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
post operative complications | 6 months
  Total number of days spent in the hospital. This will be calculated by adding the hospital length of stay for initial surgery, length of stay for any additional readmission resulting from the surgery, and emergency room visits resulting from the surgery

SECONDARY OUTCOMES:
adequacy of different techniques | 6 months to one year
  Surgical Site Infection (SSI) CDC definition
Surgical Site Occurrence (SSO) | 6 months to one year
  Hematoma, seroma, dehiscence, necrosis, non-healing wound found on abdominal exam
Hernia Reoccurence | 6 months to one year
  A hernia that was repaired in the past but has returned

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig Unversity, Zagazig, Egypt